CLINICAL TRIAL: NCT00002837
Title: Phase I-II Study of Dose Intense Doxorubicin, Paclitaxel And Cyclophosphamide With Peripheral Blood Progenitor Cells (PBPC) And Cytokine Support In Patients With Metastatic Breast Cancer
Brief Title: High-Dose Combination Chemotherapy and Peripheral Stem Cell Transplantation in Treating Patients With Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM95-156; P30CA016672 (NIH); MDA-DM-95156 (Other: UT MD Anderson Cancer Center); NCI-V96-1017; CDR0000065052 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-07-01 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Cyclophosphamide; Doxorubicin; Paclitaxel; Peripheral Blood Stem Cell Transplantation; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Doxorubicin, Paclitaxel + Cyclophosphamide with PBPC (Experimental)
  Interventions: Biological: Filgrastim (G-CSF); Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Paclitaxel; Procedure: Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: Filgrastim (G-CSF)
  Other Names: Neupogen
Drug: Cyclophosphamide
  Other Names: Cytoxan; Neosar
Drug: Doxorubicin Hydrochloride
  Other Names: Adriamycin PFS; Adriamycin RDF
Drug: Paclitaxel
  Other Names: Taxol
Procedure: Peripheral Blood Stem Cell Transplantation
  Other Names: PBSCT; Stem Cell Transplant; SCT

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining peripheral stem cell transplantation with chemotherapy may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of high-dose combination chemotherapy and peripheral stem cell transplantation in treating patients with recurrent or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Define the maximum tolerated doses of four courses of doxorubicin (DOX), paclitaxel (TAX), and cyclophosphamide (CTX) followed by peripheral blood stem cell (PBSC) and granulocyte colony-stimulating factor support given in an out-patient setting in patients with metastatic breast cancer. II. Evaluate the cardiotoxicity of the combination of bolus DOX, a 3-hour infusion of TAX, and CTX. III. Determine the clinical response rate and time to progression associated with this regimen. IV. Determine Cmax, AUC and the drug:metabolite ratio of TAX and DOX when given with CTX, a known p450 inducer.

OUTLINE: Patients without prior doxorubicin (DOX) or paclitaxel (TAX) receive two courses of induction chemotherapy with DOX/TAX with G-CSF support given 3 weeks apart. Peripheral blood stem cells (PBSC) are harvested during the recovery phase following the second course. Patients who previous received DOX or TAX and responded receive cyclophosphamide (CTX) with G-CSF for stem cell mobilization followed by PBSC harvest. Back-up bone marrow may be harvested from patients without marrow involvement for whom PBSC collection is inadequate. Patients with responding or stable disease who have adequate PBSC available receive dose-intensive chemotherapy with DOX, CTX, and TAX given on day 1, with PBSC infused on day 3 and G-CSF given from day 3 until neutrophil recovery. Four courses of dose-intensive chemotherapy with PBSC and G-CSF support are given every 3-4 weeks. During the phase I portion of the study, groups of 3-6 patients are treated at increasing doses of DOX, TAX, and CTX until the maximum tolerated dose (MTD) is determined; during the phase II portion, additional patients are treated at the MTD. Patients who progress after 2 courses of induction or 2 courses of dose-intensive chemotherapy are given the option of receiving their PBSC after conditioning with a different regimen (e.g., CTX, etoposide, and cisplatin). Patients who receive induction on protocol but who choose not to receive dose-intensive chemotherapy continue DOX/TAX for a total of 6 courses. Patients are followed 3, 6, 12, 18, and 24 months after therapy, then as clinically indicated.

PROJECTED ACCRUAL: During the phase I portion of the study, groups of 3-6 patients will be entered at each dose level studied. During the phase II portion of the study, 25 patients will be treated at the maximum tolerated dose.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed breast cancer that is metastatic or recurrent Poor-prognosis status required for Phase I portion of the study, i.e.: Estrogen receptor and progesterone receptor-negative tumor OR Failed hormonal therapy and with bulky disease or liver metastasis Bone marrow involvement less than 15% No active CNS metastases

PATIENT CHARACTERISTICS: Age: 15 to 60 Sex: Not specified Performance status: Zubrod 0 or 1 Hematopoietic: WBC greater than 3,500/mm3 Absolute granulocyte count greater than 2,000/mm3 Platelet count greater than 100,000/mm3 Hepatic: Liver function tests less than twice normal Renal: Creatinine clearance (calculated) at least 60 mL/min Cardiovascular: Left ventricular ejection fraction greater than 50% No symptomatic cardiac disease requiring antiarrhythmic or inotropic therapy Pulmonary: DLCO greater than 50% of predicted Other: No pre-existing peripheral neuropathy greater than grade 1 No severe concomitant medical or psychiatric disease

PRIOR CONCURRENT THERAPY: Biologic therapy: More than 3 weeks since any immunotherapy Chemotherapy: No prior doxorubicin or paclitaxel Patients with up to 150 mg per square meter doxorubicin or up to 4 courses of paclitaxel and who have responding disease are eligible for dose-intensive portion of protocol therapy Endocrine therapy: Not specified Radiotherapy: More than 3 weeks since any radiotherapy Surgery: Not specified

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 1995-09; Primary Completion 2002-01 (Actual); Study Completion 2002-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Doses (MTD) of 4 courses Doxorubicin, Paclitaxel, + Cyclophosphamide followed by PBSC and G-CSF Support | Evaluated with each 3-4 week course

CONTACTS AND LOCATIONS:
Overall Officials: Michele L. Donato, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org